CLINICAL TRIAL: NCT04900103
Title: Evaluation of Implementation Process of Tech-Volunteer Program in Palliative Care: ITV-Pal Program
Brief Title: Evaluation of Implementation of ITV-Pal Program
Acronym: ITV-Pal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cudeca Hospice Foundation (Other)
Collaborators: La Caixa Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SR20-00841
Record Dates: First submitted 2021-04-05; First posted 2021-05-25 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Palliative Care
Keywords: Palliative Care; Volunteering; New technologies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tech-volunteer (Experimental): A complex intervention with two phases is proposed.
  * First phase: volunteers new technologies training (tech-volunteering). Volunteers will be trained in the use of NT and their interconnectivity as tools to support their volunteer work. This training will be integrated into the PC volunteer training programme.
  * Second phase: using the NT with patients and relatives.
  Interventions: Other: ITV-Pal
- Usual volunteer (No Intervention): the control group will receive standard volunteer service.

INTERVENTIONS:
Other: ITV-Pal — Use of new technologies for volunteering
  Arms: Tech-volunteer

SUMMARY:
How can offer support to patients and families through a volunteer caring program based on new technologies? The aim of this study is to implement and evaluate a volunteer training programme in the use of new technologies: ITV-Pal Programme to support patients facing a life-threatening illness and their families.

It will created two groups of volunteers, one group will follow the CUDECA standard training program, the other will follow the proposed intervention, ITV-Pal programme. Volunteers will be allocated randomly to each group. Second stage will consist in the implementation of the direct support to patients and families through the volunteers.

The expectation is that ITV-Pal volunteers trained will be able to increase general welfare of patients and families they care for. To test it, the quality of life of patients, families and volunteers, the quality of the dying process, and identify how new technology supports volunteer end of life care will be measure.

DETAILED DESCRIPTION:
The inclusion of volunteers to the Team in the care of the patient and the family is continually increasing. The requests for volunteers by the Medical Care Teams have been increasing year after year by 5%, reaching about 75 requests received in 2019. 85% of these requests are assigned a volunteer and the 15% who are not assigned is because the volunteer does not have the required profile which responds to the patient's needs. These statistics show, on the one hand, the important and irreplaceable work that volunteers offer in social support to the patient and this is perceived both by the patient and their family who decide to have it, and also by the Care Team that is aware of the benefits of "non-professional" care, which also humanises palliative care. On the other hand, the volunteer is increasingly present in our society and this is positive, so that more people offer their collaboration and this in turn "normalises" their role in palliative care.

Although volunteers contribute millions of hours of work, the review of bibliography found no sufficiently robust studies to merit inclusion, and even less when associating PC volunteering and NT. As more research is needed on the impact of training and support for palliative care volunteers, this study intends to study the state of art of technophilia and technophobia among patients, relatives, volunteers and healthcare professionals in PC, and according to the results, implement and evaluate a volunteer training programme in the use of new technology to support patients dying at home and their relatives.

The best approach to evaluate the implementation process of complex intervention is the combination of quantitative and qualitative methods. Basic quantitative measures of implementation may be combined with in-depth qualitative data to provide detailed understandings of intervention functioning on a small scale. Use quantitative methods to measure key process variables and allow testing of pre-hypothesised mechanisms of impact and contextual moderators. Use qualitative methods to capture emerging changes in implementation, experiences of the intervention and unanticipated or complex causal pathways, and to generate new theory.

Quantitative approach:

* Pragmatic cluster randomized clinical trial to test the efficacy (the unit of randomization is the volunteer and the unit of analysis is the patient/relative).
* Before-after design for satisfaction of volunteers and HPC with the intervention and its implementation to test the effectiveness.
* Cost-utility study from the perspective of the funder with a time horizon of one year. A detailed cost analysis including costs for the adaptation of volunteer standard course to ITVPal Programme as well as the recruitment and training costs of the volunteers will be performed.

Qualitative approach: interviews (individuals and groupal) with HPC, volunteers and with key informants of patients/relatives to test at the beginning the need and usefulness of NT, and also during the implementation process to test changes and experiences.

ELIGIBILITY:
Inclusion Criteria:

Patients/relatives:

* Over 18 years; PC patients and relatives eligible for volunteer support according to the PC team assessment.
* Acceptance to participate in the study by signing the Informed Consent.

PC Volunteers:

- Acceptance to participate in the study by signing the Informed Consent.

Exclusion criteria

- No acceptance to participate in the study by signing the Informed Consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Distress thermometer | Through study completion, an average of 3 months
  Distress is an unpleasant experience of a mental, physical, social, or spiritual nature. It can affect the way you think, feel, or act. Distress may make it harder to cope with having cancer, its symptoms, or its treatment. 0 no distress 10 extreme distress
ICECAP-SCM | Through study completion, an average of 15 days
  The ICECAP Supportive Care Measure (ICECAP-SCM) has been developed as a tool for use in economic evaluation conducted in an end of life setting

SECONDARY OUTCOMES:
EuroQoL 5D-5L | Baseline, 15 and 30 days after inclusion.
  Quality of life. five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  to describe and value health across a wide range of disease areas. They are also frequently used in research into health in the general population.
Satisfaction Volunteer Programme | Through study completion, an average of 12 months
  Satisfaction with Volunteer Programme by a self develop questionaire
Service Improvement Metrics: fidelity | Through study completion, an average of 12 months
  Success of the Infrastructure. Whether the intervention was delivered as intended:
  Referral criteria/identification of patients.
Service Improvement Metrics: dose | Through study completion, an average of 12 months
  Eligibility and take up of the service. The quantity of intervention implemented: Number of patients eligible for the service and number of patients who accept the service.
Service Improvement Metrics: reach | Through study completion, an average of 12 months
  Spread of implementation. Whether the intended audience comes into contact with the intervention, and how: Number of wards with 'eligible' patients and number of wards where the service is implemented.
Heath resource use | Through study completion, an average of 12 months
  Use of health resource during the study

OTHER OUTCOMES:
PHTech questionnaire | Through study completion, an average of 3 months
  Attitudes and feelings towards technology: Technophilia/Technophobia. six items in the two factors, techEnthusiasm and techAnxiety, 1 to 5 scale so that the TechPH index could be interpreted on a five-point response scale, ranging from 1 (fully disagree) to 5 (fully agree), where the higher the index indicates a higher level of technophilia.
Volunteer Motivation (VFI) | Baseline
  A 30-item measure of motivations to volunteer. Respondents answer each item on a 7-point scale ranging from 1 (not at all important/accurate) to 7 (extremely important/accurate).
Age | Baseline
  Age of participant measured in years
Sex | Baseline
  Sex of the participant
Educational level | Baseline
  Maximun educational level completed of the participant

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación CUDECA, Benalmádena, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barnestein-Fonseca P, Vibora-Martin E, Ruiz-Torreras I, Chapinal-Bascon H, Martin-Rosello ML, Gomez-Garcia R. ITV-Pal programme: protocol of evaluation of the implementation of tech-volunteer programme in palliative care services. BMJ Open. 2023 Aug 24;13(8):e065222. doi: 10.1136/bmjopen-2022-065222. PMID 37620277